CLINICAL TRIAL: NCT04702685
Title: A Single Center, Randomized, Parallel Group Study to Evaluate the Efficacy of Ropivacaine Administered by Ultrasound-guided Erector Spinae Plane Block for Major Upper Abdominal Surgery
Brief Title: Erector Spinae Plane Block With Ropivacaine for Major Upper Abdominal Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nazarbayev University Medical Center (Other)
Collaborators: National Research Oncology and Transplantology Center, Kazakhstan (Other)
Responsible Party: Sponsor
Organization: Nazarbayev University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESP1
Record Dates: First submitted 2020-12-03; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Pain, Postoperative
Keywords: ropivacaine; major upper abdominal surgery; supraumbilical; liver resection; colon resection; Whipple procedure; gastrectomy; anesthetics, local; erector spinae plane block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Bandage with tape will be placed over the presumed site of anesthetic injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine (Experimental): Ropivacaine 0.5% - 20 ml will be administered as erector spinae plane block under ultrasound guidance
  Interventions: Drug: Ropivacaine
- Placebo (Placebo Comparator): No injection. Bandage will be placed over the presumed site of injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ropivacaine — Local anesthetic for injection
  Other Names: Naropin
  Arms: Ropivacaine
Other: Placebo — Bandage will be placed in the presumed injection site while patients in under general anesthesia
  Arms: Placebo

SUMMARY:
Prospective, single-centre, randomized, controlled, open-label, evaluator-blinded, superiority trial.

DETAILED DESCRIPTION:
The primary objective is to establish whether ESP ropivacaine reduces post-operative opioid use and improves pain rating post-operatively. The secondary objectives include adverse event incidence, time to ambulation and time to discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Adults who are scheduled to undergo major upper abdominal surgery (e.g. Pancreato-duodenal resection). If enrollment rates are insufficient, patients undergoing other major upper abdominal surgery will be enrolled (e.g in the supraumbilical area: liver resection, colon resection; Whipple procedure; gastrectomy).
2. Males or females 18-70 years of age
3. American Society of Anesthesiologists physical status class I,II, III
4. Signed informed consent

Exclusion Criteria:

1. Patients undergoing emergency surgery
2. Decompensated cardiovascular disease (e.g. left ventricular ejection fraction ≤40%), chronic heart failure, rhythm and conduction disorders, coagulopathies)
3. Comorbid obesity (BMI≥35kg/m2)
4. Anomalies of vertebral column
5. Use of anticoagulants and patients with hypocoagulable conditions
6. Pregnancy
7. Physician preference for therapeutic anticoagulation
8. Infection of skin at site of needle puncture
9. Known allergies to study drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Mean cumulative opioid consumption up to 24 hours after surgery | 24 hours post-operation
  Cumulative opioid consumption will be recorded for 24 hours following surgery

SECONDARY OUTCOMES:
Post-operative pain score | Measured post-operatively at 0, 2, 4, 6, 8, 10, 12, 16, 20, 24 hours after surgery.
  Numerical rating scale (0= no pain; 10= worst pain imaginable) will be used
Time to ambulation | Between surgery and discharge from hospital, expected time is between 1 day to 1 week
  The time that the patient is able to walk independently, after surgery
Time to discharge | Expected time to discharge is up to 2 weeks
  From time of surgery completion to discharge from hospital
Usage of NSAIDs post surgery | Total dose used during the 24 hour period after surgery.
  Dose

CONTACTS AND LOCATIONS:
Overall Officials: Philip la Fleur, RPh MSc, Principal Investigator — philip.lafleur@nu.edu.kz
Locations (1):
- National Center for Oncology, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
Upon request, we will share information with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Q3 and Q4 2021
Access Criteria: Researchers on staff at an accredited university